CLINICAL TRIAL: NCT03262272
Title: Evaluation of Dialyzers' Biocompatibility and Performances Compared in Different Dialysis Treatments : Conventional Hemodialysis and Post-dilution Hemodialfiltration
Brief Title: Evaluation of Biocompatibility and Performances of 4 Dialyzers in Different Mode Treatments
Acronym: BIOMODAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hemotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIOMODAL 2016-A01122-49
Record Dates: First submitted 2017-07-12; First posted 2017-08-25 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: End Stage Renal Disease; Inflammation
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation

STUDY DESIGN:
Intervention Model Description: Prospective randomized cross-over study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodialysis (Experimental): patients treated by conventionnal hemodialysis
  Interventions: Device: VIE A Hemodialyzer; Device: Rexsys 27H hemodialyzer; Device: Leoceed 21HX hemodialyzer; Device: Polypure 22S+ hemodialyzer
- Hemodiafiltration post dilution (Experimental): patients treated by HDF post-dilution
  Interventions: Device: VIE A Hemodialyzer; Device: Rexsys 27H hemodialyzer; Device: Leoceed 21HX hemodialyzer; Device: Polypure 22S+ hemodialyzer

INTERVENTIONS:
Device: VIE A Hemodialyzer — polysulfon membrane coated with vitamin E
Device: Rexsys 27H hemodialyzer — polyethersulfon membrane with large surface area : 2,7m²
Device: Leoceed 21HX hemodialyzer — polyslfon membrane with gamma sterilization
Device: Polypure 22S+ hemodialyzer — polysulfon membrane with steam sterilization

SUMMARY:
Prospective multicenter randomized cross-over study Number of patients : 32 (8 patients per group) Obtain objectives data to advise each hemodialyzer according to dialysis treatment and patient profile.

To evaluate the different hemodialyzers and judge their extraction performances in HD and post HDF.

Evaluation of the biocompatibility of the hemodialyzers and the patients' inflammatory status.

DETAILED DESCRIPTION:
Medical devices studied :

* Leoceed 21HX, hemodialyzer, High permeability PS membrane 2,1 m² , made by Nx Stage in Germany
* Polypure 22S, hemodialyzer, High permeability PS membrane 2,2 m² , made by Allmed in Germany
* VIE 21A hemodialyzer, High permeability PS membrane 2,1 m² coated in vitamin E, made by Asahi Kasei Medical in Japan
* Rexsys 27H, hemodialyzer , High permeability PES membrane 2,7 m² , made by Medica in Italia

These hemodialyzers are EC marked and are used in their own indications.

Schema

Details of the cross-over plan :

8 patients will be treated successively with the 4 hemodialyzers. Patients will be treated with the dialyzer "test" for the two first sessions of the week. During the last dialysis session of each week, only their usual dialyzer will be used as wash-out. A randomization will define the order of use of the dialyzers in the 4 centers. This order will be identical in a center.

Number of patients :

32 (8 patients per center (4 centers))

Duration :

One week per dialyzer

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with chronic kidney disease dialyzed for at least one month and treated with the treatment mode that we will test
* Patient using post-dilution HDF mode have to use EuDIAL volume guidelines (20-22L minimum)
* Patient treated before with high permeability membrane
* Patient with vascular access allowing a blood flow rate with a minimum of 300 mL/min
* Patient treated with a high surface area dialyzer ≥ 1,8 m²
* Patient covered by the social French health organism
* Patient informed of the study goals and having signed the informed consent

Exclusion Criteria:

* Patient with a vascular access not allowing a blood flow rate minimum of 300 mL/min
* Patient with a fast progressive chronic disease
* Patient with an uncontrolled anemia
* Patient refusing to sign the informed consent
* Pregnant or nursing patient
* Pediatric patient
* Patient under tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of middle molecules extraction | one week per dialyzer per patient
  Measurements of β 2 microglobulin (11,8kDa), myoglobin (17kDa), Beta Trace (21kDa), Free immunoglobulin light chains Kappa (23kDa), myostatin (40kDa), glycoprotein orosomucoïd (44kDa)

SECONDARY OUTCOMES:
Extraction of uremic toxins | one week per dialyzer per patient
  * Urea
  * Creatinin
  * inorganic phosphates
Biocompatibility assessment | one week per dialyzer per patient
  * Anaphylatoxins (C3a, C5a) during the session (T0, T15, Tend)
  * TNF-α and IL-6 (T0 et Tend)
Monitoring of Nutrition status | one week per dialyzer per patient
  Quantification of the albumin loss in the used dialysate (1 center) during the middle session of the week for each dialyzer tested per patient, i.e 4 times/patient.
  2 analysis modalities will be used: " pull and push " syringe Plastipak BD 50mL or collection of the whole dialysate in a 200 L tank
  Dosage Albumin et pre-albumin before dialysis session
Handling of the devices | one week per dialyzer per patient
  - Evaluation of the priming and recovery for each dialysis session
Dialysis adequacy evaluation | one week per dialyzer per patient
  Calculation of KT/V
Session tolerance | one week per dialyzer per patient
  All secondary troubles will be noted: cramps, nauseas, hypotension…
Parameters inflammation | one week per dialyzer per patient
  CRP (mg/l)
Parameters inflammation | one week per dialyzer per patient
  - Calcul of PINI = [CRP(mg/l) x Orosomucoïd (mg/l)] / [Albumin(g/l) x Pre-albumin(mg/l)]

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul CRISTOL, Professor, Study Director — University Hospital, Montpellier
Locations (1):
- AIDER-Lapeyronie, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kokubo K, Kurihara Y, Kobayashi K, Tsukao H, Kobayashi H. Evaluation of the Biocompatibility of Dialysis Membranes. Blood Purif. 2015;40(4):293-7. doi: 10.1159/000441576. Epub 2015 Nov 17. PMID 26656534
- [Background] Maduell F, Moreso F, Mora-Macia J, Pons M, Ramos R, Carreras J, Soler J, Torres F; study group ESHOL. ESHOL study reanalysis: All-cause mortality considered by competing risks and time-dependent covariates for renal transplantation. Nefrologia. 2016;36(2):156-63. doi: 10.1016/j.nefro.2015.10.007. Epub 2015 Dec 8. English, Spanish. PMID 26672890